CLINICAL TRIAL: NCT03036410
Title: Evaluation of Different Phone Solutions in CI and Hearing Aid Users and Bimodal Recipients
Acronym: PhoneCIHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics AG (Industry)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AK-KEK-2016-01853
Record Dates: First submitted 2017-01-16; First posted 2017-01-30 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Hearing Loss, Binaural; Hearing Loss, Monaural
Keywords: Hearing Aid Usage (monaural, binaural); Cochlear Implant Usage (monaural, binaural); Hearing Aid and Cochlear Implant Usage (monaural)
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bimodal user (Other): wearing one hearing aid and one CI Intervention: Standard Phone, DECT Phone, Easy Call, Duo Phone
  Interventions: Device: standard telephone setting; Device: DECT; Device: EasyCall; Device: DuoPhone
- unilateral hearing aid users (Other): wearing one hearing aid Intervention: Standard Phone, DECT Phone, Easy Call, Duo Phone
  Interventions: Device: standard telephone setting; Device: DECT; Device: EasyCall
- bilateral hearing aid users (Other): wearing two hearing aids Intervention: Standard Phone, DECT Phone, Easy Call, Duo Phone
  Interventions: Device: standard telephone setting; Device: DECT; Device: EasyCall; Device: DuoPhone
- CI users (Other): wearing CI Intervention: Standard Phone, DECT Phone, Easy Call, Duo Phone
  Interventions: Device: standard telephone setting; Device: DECT; Device: EasyCall; Device: DuoPhone

INTERVENTIONS:
Device: standard telephone setting — without streaming function
Device: DECT — cordless telephone (streaming to both hearing devices)
Device: EasyCall — accessories for Bluetooth capable mobile telephones (streaming to both hearing devices)
Device: DuoPhone — streaming function, which provides the speech signal to both ears
  Arms: CI users; bilateral hearing aid users; bimodal user

SUMMARY:
Communication on telephone is challenging for people with hearing loss. For hearing aid users, for instance, the inventions for improving speech intelligibility on the phone range from an integrated tele coil and individual hearing programs to specially designed phone devices. No formal studies involving these devices have been carried out with CI users.

Thus, this comparative study includes hearing aid as well as CI and bimodal users to evaluate different hearing solutions for communication on telephone in terms of intelligibility and ease of use.

DETAILED DESCRIPTION:
Communication on telephone is challenging for people with hearing loss, due to a number of factors:

* The lack of visual cues (lip-reading),
* The lack of binaural abilities,
* The presence of (loud) background noise in a variety of listening situations,
* A modified speech signal due to reduced frequency bandwidth and
* Difficulties coupling the phone to the CI. For hearing aid users, for instance, the inventions for improving speech intelligibility on the phone range from an integrated tele coil and individual hearing programs to specially designed phone devices.

No formal studies involving these devices have been carried out with CI users.

Thus, this comparative study includes hearing aid as well as CI and bimodal users to evaluate the different hearing solutions for communication on telephone in terms of intelligibility and ease of use:

* Phonak DECT - cordless telephone for HA-, CI- users and bimodal users
* Phonak EasyCall - accessories for Bluetooth capable mobile telephones for HA-, CI- and bimodal users
* Phonak DuoPhone - streaming function, which provides the speech signal to both ears

ELIGIBILITY:
Inclusion Criteria:

* Unilateral HA users with SRT of better (lower) than + 3 dB
* Bilateral HA users with SRT of better (lower) than 0 dB
* Unilateral CI users:

Unilaterally implanted with an Advanced Bionics CII, HiRes90k or Advantage implant

1-year acclimatization time after implantation at least 20% correct for a sentence test delivered with a SNR of + 10 dB, or a SRT of better (lower) than + 15 dB

* Bimodal (CI + HA) users:

Unilaterally implanted with an Advanced Bionics CII, HiRes90k or Advantage implant CI side: at least 20% correct for a sentence test delivered with a SNR of + 10 dB, or a SRT of better (lower) than + 15 dB HA side: unaided threshold ≤ 80 dB at least for frequencies up to 500 Hz

* All users:

Informed Consent as documented by signature Ability for speech understanding in the presence of competing noise without any assistance from lip-reading Ability to give subjective feedback in a certain listening situation First language: German or Swiss-German

Exclusion Criteria:

* All users:

Difficulties additional to hearing impairment that would interfere with the study procedures Acute inflammation or pain in head-/neck area Dizziness Age of participants < 18 years Age of participants > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
speech reception threshold (SRT) assessment with audiological measures | 6 months
  differences in speech reception threshold (SRT) on the phone in the presence of background noise between the Phonak DECT phone and a standard phone will be assessed with audiological measures.

SECONDARY OUTCOMES:
Subjective ratings assessment with scaling | 6 months
  * differences in preference ratings in the presence of background noise between a standard phone, a standard phone + DuoPhone algorithm, the DECT-telephone
  * differences in preference ratings in the presence of background noise between a standard mobile phone, a standard mobile phone + DuoPhone algorithm and a standard mobile phone + EasyCall accessory

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Department of Otorhinolaryngology, Head and Neck Surgery, Zurich, Switzerland

REFERENCES:
- [Background] Cray JW, Allen RL, Stuart A, Hudson S, Layman E, Givens GD. An investigation of telephone use among cochlear implant recipients. Am J Audiol. 2004 Dec;13(2):200-12. doi: 10.1044/1059-0889(2004/025). PMID 15903146
- [Background] Anderson I, Baumgartner WD, Boheim K, Nahler A, Arnoldner C, D'Haese P. Telephone use: what benefit do cochlear implant users receive? Int J Audiol. 2006 Aug;45(8):446-53. doi: 10.1080/14992020600690969. PMID 17005487
- [Background] Adams JS, Hasenstab MS, Pippin GW, Sismanis A. Telephone use and understanding in patients with cochlear implants. Ear Nose Throat J. 2004 Feb;83(2):96, 99-100, 102-3. PMID 15008443
- [Background] Picou EM, Ricketts TA. Comparison of wireless and acoustic hearing aid-based telephone listening strategies. Ear Hear. 2011 Mar-Apr;32(2):209-20. doi: 10.1097/AUD.0b013e3181f53737. PMID 20808225
- [Background] Picou EM, Ricketts TA. Efficacy of hearing-aid based telephone strategies for listeners with moderate-to-severe hearing loss. J Am Acad Audiol. 2013 Jan;24(1):59-70. doi: 10.3766/jaaa.24.1.7. PMID 23231817